CLINICAL TRIAL: NCT04935424
Title: Evaluation of Treatment for Leukoderma by Cellular Level Resolution Full-field Optical Coherence Tomography
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Apollo Medical Optics, Ltd (Industry)
Responsible Party: Principal Investigator, Chau Yee Ng, Principal Investigator, Chang Gung Memorial Hospital
Other Study IDs: 20STW2-4-010-V1A3
Record Dates: First submitted 2021-05-04; First posted 2021-06-23 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Leukoderma
Keywords: Optical coherence tomography (OCT); dermatology; Full-Field OCT; Non-invasive image system; Leukoderma
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental：Leukoderma: Device: ApolloVue® S100 image system
  Interventions: Device: ApolloVue® S100 Image System (Apollo Medical Optics)

INTERVENTIONS:
Device: ApolloVue® S100 Image System (Apollo Medical Optics) — The device is an in vivo non-invasive optical coherence tomography and will be used to obtain at least 6 medical images of normal and lesional skin, respectively, for both experimental group and control group. The ApolloVue S100 image system is a high resolution OCT imaging system that provide real-time visualization of human skin tissue microstructure. The system provides cellular level, two-dimensional, cross-sectional (B-scan) and en face (E-scan) that can assist clinical diagnosis.The system is also equipped with imaging guiding system that could assist in position scanning skin area.
  Other Names: 510(K) Number: K201552 (class II)

SUMMARY:
OCT is an optical technology that emerged as a non-invasive skin imaging for the skin. In this protocol, the investigators plan to study the optical imaging features of leukoderma. An estimated 65 subjects will be included in this trial.

This is an observational, non-randomised, non-controlled, prospective cohort study to observe the feasibility of in vivo OCT as a image tool in the diagnosis of leukoderma. Use of the device will not affect the clinical management of the subjects.

Scientific Aim:

To evaluate the feasibility ApolloVue S100 image system as a tool in the differential diagnosis of leukoderma..

ELIGIBILITY:
Inclusion Criteria:

1. Age ≧ 20
2. Subject with at least one leukoderma lesion
3. Willing to participate in the trial with informed consent

Exclusion Criteria:

1. Age < 20
2. Pregnant woman or woman wishing to be pregnant during the study, or during breastfeeding period
3. The investigators consider inappropriate to participate in the trial.
4. Open wound lesion.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject with at least one leukoderma lesion
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
To describe characteristic features seen by Full-field Optical Coherence Tomography of leukoderma disorders. | 6 months
  The study is a descriptive one. To researche the characteristic images of leukoderma. No formal statistical testing of correlations will be performed. All images will be evaluated as a group. First, the investigator will review the OCT images for each imaging site and will determine the presence/absence of leukoderma. Next, comparing with the leukoderma disorders images to highlight any features that may assist in the OCT evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu Z, Jiang M, Zhao J, Wang Q, Zhang C, Gao M, Gu M, Xiang L. Efficacy of a wound-dressing biomaterial on prevention of postinflammatory hyperpigmentation after suction blister epidermal grafting in stable vitiligo patients: a controlled assessor-blinded clinical study with in vitro bioactivity investigation. Arch Dermatol Res. 2020 Nov;312(9):635-645. doi: 10.1007/s00403-020-02049-2. Epub 2020 Feb 27. PMID 32107629
- [Background] Abdel-Malek ZA, Jordan C, Ho T, Upadhyay PR, Fleischer A, Hamzavi I. The enigma and challenges of vitiligo pathophysiology and treatment. Pigment Cell Melanoma Res. 2020 Nov;33(6):778-787. doi: 10.1111/pcmr.12878. Epub 2020 Apr 12. PMID 32198977
- [Background] Li W, Wang S, Xu AE. Role of in vivo reflectance confocal microscopy in determining stability in vitiligo: a preliminary study. Indian J Dermatol. 2013 Nov;58(6):429-32. doi: 10.4103/0019-5154.119948. PMID 24249892
- [Background] Alghamdi KM, Kumar A, Taieb A, Ezzedine K. Assessment methods for the evaluation of vitiligo. J Eur Acad Dermatol Venereol. 2012 Dec;26(12):1463-71. doi: 10.1111/j.1468-3083.2012.04505.x. Epub 2012 Mar 15. PMID 22416879
- [Background] Kang HY, Bahadoran P, Ortonne JP. Reflectance confocal microscopy for pigmentary disorders. Exp Dermatol. 2010 Mar;19(3):233-9. doi: 10.1111/j.1600-0625.2009.00983.x. Epub 2009 Nov 2. PMID 19889023
- [Background] Lai LG, Xu AE. In vivo reflectance confocal microscopy imaging of vitiligo, nevus depigmentosus and nevus anemicus. Skin Res Technol. 2011 Nov;17(4):404-10. doi: 10.1111/j.1600-0846.2011.00521.x. Epub 2011 Mar 24. PMID 21429011